CLINICAL TRIAL: NCT05094362
Title: Operant Conditioning of Spinal Reflexes to Enhance Motor Function Recovery After Spinal Cord Injury
Brief Title: Operant Conditioning of Spinal Reflexes Training System--Reflex Operant Down Conditioning
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of South Carolina (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Aiko Thompson, Associate Professor, Medical University of South Carolina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00095583; 4U44NS114420-03 (NIH)
Record Dates: First submitted 2021-10-14; First posted 2021-10-26 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord Injuries; Neurological Injury; Paralysis; Spasticity, Muscle
Keywords: Neuroplasticity; Spinal Reflex
MeSH Terms: conditions — Spinal Cord Injuries; Trauma, Nervous System; Paralysis; Muscle Spasticity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Validation of the new training system (Experimental): The researchers will measure changes in H-reflex size achieved with the use of the new system and compare these measures with the existing results in 25 spastic individuals with chronic incomplete SCI. Each participant completes 6 baseline sessions and 30 conditioning sessions. In the 30 conditioning sessions, the soleus H-reflex will be down-conditioned to decrease the activity of the hyperactive spinal stretch reflex pathway in people with spasticity that is characterized by exaggerated reflex activity. It is anticipated that the magnitude of reflex change obtained with the use of the new system would be greater or at least the same as the bench-marked values from the previous studies that used the old prototype reflex conditioning system.
  Interventions: Behavioral: Spinal Reflex Operant Down Conditioning

INTERVENTIONS:
Behavioral: Spinal Reflex Operant Down Conditioning — This is a training intervention in which people with a spinal cord injury are trained to reduce the activity of a certain spinal reflex. By decreasing this reflex, individuals decrease hyperactivity in the reflex and can reduce spasticity.

SUMMARY:
The purpose of this study is to validate the capacity of a reflex training system to change the size of the targeted reflex. For this, the researchers are recruiting 25 individuals with chronic incomplete SCI who have spasticity in the leg to participate in the reflex training procedure. The study involves approximately 45 visits with a total study duration of about 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. a clinically stable spinal cord injury (above T11) that occurred at least one year previously
2. the ability to ambulate at least 10 m with or without an assistive device (i.e., walker, crutches, or cane, not parallel bars) within 100 sec (those with 10-meter walking time >100 sec are excluded because it is unlikely that they are able to participate in and complete our planned locomotion evaluation procedures)
3. clinical signs of spasticity in the plantarflexor muscles at least unilaterally (i.e., hyperreactivity to Achilles tendon tap, and increased muscle tone, score >1 on Modified Ashworth scale)
4. spastic hyperreflexia reflected in exaggerated H-reflex
5. functionally and medically stable for at least 3 months
6. medical clearance to participate
7. reasonable expectation that current medications (including antispasticity medication such as baclofen, diazepam, and tizanidine) will not change over the conditioning period. Each participant's medication and dosage will be monitored and recorded throughout the study. Once enrolled, the subject will remain enrolled even if medication changes. (Because only neurologically stable subjects will enter this study, medication changes will be unlikely.)

Exclusion Criteria:

1. motoneuron injury;
2. a cardiac condition (history of myocardial infarct, pacemaker use, etc.)
3. an unstable medical condition
4. a pre-existing or confounding neurological condition (e.g., history of Multiple Sclerosis (MS), Traumatic Brain Injury (TBI), Stroke, Parkinson's disease)
5. a condition that prevents lower extremity mobility testing or weight bearing (e.g. fracture, severe sprain/strain, botox muscular injection) (orthotic knee hyperextension is not excluded; in severe cases of knee hyperextension, the brace can be worn during the study sessions)
6. a cognitive impairment that precludes giving informed consent (e.g., severe intellectual disability)
7. use of a functional electrical stimulation (FES) foot-drop stimulator or an FES bicycle on a daily basis (FES applied to the arm is acceptable)
8. deep vein thrombosis within the past 6 months
9. depression (due to potential interference of anti-depressant medication with the intervention and possible reduced participation reliability)
10. pregnancy (due to expected changes in weight and posture and potentially unstable medical condition).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2023-08-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in reflex activity as measured by the H-reflex amplitude (mV) in response to nerve stimulation | Before Baseline, after completion of intervention sessions (approximately 10 weeks), 1 month and 3 months after the completion of intervention
  Decreased H-reflex amplitude indicates reduced reflex activity and a more normal reflex response to muscle activity
Change in walking speed (m/s) as measured by the 10-meter Walk Test (10MWT) | Before Baseline, after completion of intervention sessions (approximately 10 weeks), 1 month and 3 months after the completion of intervention
  Speed of the participant's fastest comfortable walking speed across 10 meters. Decreased time (sec) demonstrates increased walking speed (m/s)
Change in walking distance (meters) as measured by the 6-minute walk test | Before Baseline, after completion of intervention sessions (approximately 10 weeks), 1 month and 3 months after the completion of intervention
  The distance walked in 6 minutes in measured. The participant is asked to walk at his/her fastest comfortable speed on an indoor walkway.

SECONDARY OUTCOMES:
Change in the level of assistance required to walk 10 meters as measured by the Walking Index for Spinal Cord Injury (WI-SCI) | Before Baseline, after completion of intervention sessions (approximately 10 weeks), 1 month and 3 months after the completion of intervention
  WI-SCI classifies the level of assistance needed to perform the 10MWT; the scale is from 0-20 with 20 being no assistance required at all. An increase of score indicates increased level of independence while walking.
Change in level of spasticity in the more affected leg as measured by the Modified Ashworth Scale (MAS) | Before Baseline, after completion of intervention sessions (approximately 10 weeks), 1 month and 3 months after the completion of intervention
  A decrease in the score on the MAS indicates a decrease in spasticity. To measure spasticity, resistance to passive movement about a joint is tested at a range of velocities. The score ranges from 0-4 (i.e., 0: normal muscle tone; 4: rigid in flexion or extension).
Change in balance as measured by Berg Balance Scale | Before Baseline, after completion of intervention sessions (approximately 10 weeks), 1 month and 3 months after the completion of intervention
  An increase in score on the Berg Balance scale indicates better balance and decreased fall risk. For each item, the score ranges from 0-4 with a maximum total score of 56.
Change in basic functional independence as measured by the Spinal Cord Independence Measure (SCIM III) | Before Baseline, after completion of intervention sessions (approximately 10 weeks), 1 month and 3 months after the completion of intervention
  An increase in the the score on the SCIM III indicates increased basic functional independence. This is a self report questionnaire with 19 items in three sub-scales: (1) self-care (6 items, subscore 0-20); (2) respiration and sphincter management (4 items, subscore 0-40); and (3) mobility (9 items, subscore 0-40). The total score ranges from 0-100.
Change in functional independence as measured by the Functional Independence Measure (FIM) | Before Baseline, after completion of intervention sessions (approximately 10 weeks), 1 month and 3 months after the completion of intervention
  An increase in the score on the FIM indicates and increase in functional independence. This 18-item, clinician-reported scale assesses function in 6 areas including self-care, continence, mobility, transfers, communication, and cognition. Each of the 18 items is graded on a scale of 1-7 based on level of independence in that item (1 = total assistance required, 7 = complete independence).
Change in quality of life as measured by Spinal Cord Injury Quality of Life and Participation Questionnaire (SCI-QOL) | Before Baseline, after completion of intervention sessions (approximately 10 weeks), 1 month and 3 months after the completion of intervention
  An increase in score on the SCI-QOL indicates an increase in quality of life.
Change is strength of key muscles in the lower extremity as measured by Manual Muscle Testing (MMT) | Before Baseline, after completion of intervention sessions (approximately 10 weeks), 1 month and 3 months after the completion of intervention
  To test the strength against the examiner's resistance and grading the patient's strength on a 0 to 5 scale. 0: No muscle activation; 1: Trace muscle activation, such as a twitch, without achieving full range of motion; 2: Muscle activation with gravity eliminated, achieving full range of motion; 3: Muscle activation against gravity, full range of motion; 4: Muscle activation against some resistance, full range of motion; 5: Muscle activation against examiner's full resistance, full range of motion.
Change in dynamic and static muscle length and joint range of motion (ROM) as measured by Tardieu Scale | Before Baseline, after completion of intervention sessions (approximately 10 weeks), 1 month and 3 months after the completion of intervention
  An increase in joint range of motion (deg) indicates ROM more similar to individuals without injury

CONTACTS AND LOCATIONS:
Overall Officials: Aiko Thompson, PhD, Principal Investigator — Medical University of South Carolina
Locations (1):
- Medical University of South Carolina, Charleston, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No